CLINICAL TRIAL: NCT02817204
Title: Effect of Aerobic EXercise on MiCroVAscular RarefacTION in Chinese Mild HyperteNsive Patients（EXCAVATION-CHN1）
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Jun Tao, Professor,PhD, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HVD001
Record Dates: First submitted 2016-06-22; First posted 2016-06-29 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Primary Hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aerobic Exercise group (Experimental): Cardio Pulmonary Exercise Test(CPET) Cycle ergometer exercise for 3 sessions a day (3 minutes Warm up,45 minutes Resistance Exercise at 75% of HRmax;10 minutes Recovery). 5 days a week(about 2000kcal) and continues 12 weeks
  Interventions: Behavioral: Aerobic Exercise; Behavioral: Health Education
- Health Education Group (Other): Lower salt,fat and calorie diet,Recommendation of regular exercise,No smoking and alcohol Cardio Pulmonary Exercise Test(CPET) No Cycle ergometer exercise
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Behavioral: Aerobic Exercise — Cycle ergometer exercise for 3 sessions a day (3 minutes Warm up,45 minutes Resistance Exercise at 75% of HRmax;10 minutes Recovery). 5 days a week(about 2000kcal) and continues 12 weeks
  Arms: Aerobic Exercise group
Behavioral: Health Education — Lower salt,fat and calorie diet,Recommendation of regular exercise,No smoking and alcohol

SUMMARY:
The purpose of this study is to determine the effect of aerobic exercise training on microcirculation rarefaction in Chinese young male primary hypertensive patients stage 1. Hypertension is one of the most common world-wide chronic diseases, and it is showing a growing younger trend, which with mild blood pressure elevated would not be diagnose in time until blood pressure raises up or symptoms show up (Mild blood pressure indicates blood pressures ranging from 140 to 159 mmHg systolic and/or 90 to 99 mmHg diastolic). However, cumulative evidences prove that microvascular rarefaction exist in hypertensive patients with even primary hypertension stage 1. Exercise prescription is gathering great importance in preventive health. Aerobic exercise, especially, has the potential to diminish blood pressure values, and aerobic exercise can promote angiogenesis in coronary heart disease. Notch signaling plays an important role in vascular formation and maintenance. However, there is no prospective, randomized, controlled, clinic trial to investigate the effect of exercise on microcirculation rarefaction in hypertension. In summary, investigators propose a hypothesis that aerobic exercise might not only have a blood pressure lowing effect but also improve microcirculation rarefaction in Chinese male adults with primary mild hypertension. For that, subjects will be enrolled for one pre-intervention cardiopulmonary exercise test (CPET) and then randomized in aerobic exercise intervention group and control group (only health education), the intervention will be carried out by Cycle Ergometer, the protocol consists of 3 sessions a day: 3 minutes Warm up, 45 minutes Resistance Exercise at 75% of HRmax; 10 minutes Recovery. Thus 58 minutes a day and 5 days a week (about 2000kcal) and 12 weeks in total. Prior and after all intervention sessions (12 weeks), nail fold capillary microscopy and retinal capillary Optical Coherence Tomography(OCT) angiography will be assessed, as well as 24h blood pressure monitoring, echocardiography, forearm blood flow and reactive hyperemia by venous occlusion plethysmography (FMD), PWV, central arterial pressure, RHI with Endopat, also the quantification of endothelial progenistor cells(EPCs) separated from peripheral blood.

DETAILED DESCRIPTION:
Hypertension is one of the most common world-wide chronic diseases, and it is showing a growing younger trend, which with mild blood pressure elevated would not be diagnose in time until blood pressure raises up or symptoms show up (Mild blood pressure indicates blood pressures ranging from 140 to 159 mmHg systolic and/or 90 to 99 mmHg diastolic). However, cumulative evidences prove that microvascular rarefaction exist in hypertensive patients with even primary hypertension stage 1. Exercise prescription is gathering great importance in preventive health. Aerobic exercise, especially, has the potential to diminish blood pressure values, and aerobic exercise can promote angiogenesis in coronary heart disease. Notch signaling plays an important role in vascular formation and maintenance. However, there is no prospective, randomized, controlled, clinic trial to investigate the effect of exercise on microcirculation rarefaction in hypertension. In summary, investigators propose a hypothesis that aerobic exercise might not only have a blood pressure lowing effect but also improve microcirculation rarefaction in Chinese male adults with primary mild hypertension. For that, subjects will be enrolled for one pre-intervention cardiopulmonary exercise test (CPET) and then randomized in aerobic exercise intervention group and control group (only health education), the intervention will be carried out by Cycle Ergometer, the protocol consists of 3 sessions a day: 3 minutes Warm up, 45 minutes Resistance Exercise at 75% of HRmax; 10 minutes Recovery. Thus 58 minutes a day and 5 days a week (about 2000kcal) and 12 weeks in total. Prior and after all intervention sessions (12 weeks), nail fold capillary microscopy and retinal capillary Optical Coherence Tomography(OCT) angiography will be assessed, as well as 24h blood pressure monitoring, echocardiography, forearm blood Flow Mediated Diastolic function(FMD), Plus Wave Velocity(PWV), Reactive Hyperemia Index(RHI) with Endopat, also the quantification of endothelial progenistor cells(EPCs) separated from peripheral blood.

ELIGIBILITY:
Inclusion Criteria:

* Subjects range from 18 to 40 years old.
* male
* Blood pressure is primary hypertension stage I(systolic blood pressure 140 to 159 mmHg and/or diastolic blood pressure 90 to 99 mmHg).
* Able to participate in exercise
* No regular physically active in the last 4 months
* Provide informed consent and willingness to cooperate with the study protocol

Exclusion Criteria:

* Less than 18 years old or above 40 years old
* Secondary hypertension.
* Females
* Systemic diseases such as diabetes, HIV/AIDS, liver disease, chronic renal failure, tuberculosis, and autoimmune diseases
* Medical history of cardiovascular disease: acute myocardial infarct, stable angina, unstable angina, heart failure, atrial fibrillation, atrioventricular blockade, peripheral vascular disease or cerebrovascular accident
* Patients who are unfavorable of long-term follow-up or poor compliance

Ages: 25 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-07-30 (Estimated); Study Completion 2017-07-30 (Estimated)

PRIMARY OUTCOMES:
Retinal capillary density with Quantitative Optical Coherence Tomography(OCT) angiography(OCT)) | Change from Baseline retinal capillary density at 12 weeks
Nail fold capillary numbers per square millimeter( /mm²) | Change from Baseline nail fold capillary density at 12 weeks

SECONDARY OUTCOMES:
24 hours ambulatory blood pressure (ABP) in millimeters of mercury(mmHg) | Change from Baseline Systolic Blood Pressure and Diastolic Blood Pressure at 12 weeks
Flow-mediated Dilation(FMD) in % | Change from Baseline percentage at 12 weeks
  The percentage change in brachial artery diameter from baseline
Reactive Hyperemia Index(RHI) in the ratio of the average amplitude of the PAT signal | Change from Baseline ratio at 12 weeks
  RHI was measured using the RH-PAT system (EndoPAT):A blood pressure cuff was placed on 1 upper arm with the contralateral arm serving as a control. A PAT probe was placed on 1 finger of each hand. After a 5-minute equilibration period, the cuff was inflated to 60 mm Hg above the systolic pressure or to 200 mm Hg for 5 minutes, then deflated to induce reactive hyperemia.
Abilities of tube formation of endothelial progenistor cells(EPCs) in tube numbers | Change from Baseline tube numbers at 12 weeks
  Tube formation ability of EPCs was evaluated by counting tube numbers. Images of tube morphology were taken under the inverted phase contrast microscope.
Left Ventricular End-diastolic Volume (LVEDV) in milliliter(ml) | Change from Baseline volume at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Haipeng Xiao, PhD, Study Chair — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- First Affiliated Hospital,Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liang J, Li Y, Chen L, Xia W, Wu G, Tong X, Su C, He J, Lin X, Tao J. Systemic microvascular rarefaction is correlated with dysfunction of late endothelial progenitor cells in mild hypertension: a substudy of EXCAVATION-CHN1. J Transl Med. 2019 Nov 12;17(1):368. doi: 10.1186/s12967-019-2108-8. PMID 31718666